CLINICAL TRIAL: NCT00679263
Title: A Randomized, Single-blind, Parallel Group, Placebo-controlled, Dose Rate Escalation Study Evaluating the Safety and Effects of MN-221 in Subjects Diagnosed With Moderate to Severe Asthma
Brief Title: Study Evaluating the Safety and Effects of MN-221 in Subjects With Moderate to Severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediciNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MN-221-CL-005
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Results first posted 2011-12-15 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-11

CONDITIONS: Asthma
Keywords: asthma; randomized; placebo controlled; dose escalation; safety; efficacy; single blind; MN-221
MeSH Terms: conditions — Asthma | interventions — bedoradrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- MN-221 (Experimental)
  Interventions: Drug: MN-221
- PLACEBO (Placebo Comparator): Placebo intravenous infusion with dosing volume equivalent to active treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MN-221 — Initial dose: 16 μg/min for 15 minutes followed by 8 μg/min for 105 minutes (2-hour infusion with a total dose of 1,080 μg)
  Arms: MN-221
Drug: MN-221 — Subsequent dose: 30 μg/min for 15 minutes followed by 15 μg/min for 45 minutes (1-hr infusion with a total dose of 1,125 μg).
  Arms: MN-221
Drug: Placebo — Placebo intravenous infusion with dosing volume equivalent to active treatment.
  Arms: PLACEBO

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of MN-221 at two different dosing rates administered through a continuous infusion in subjects diagnosed with moderate to severe asthma.

DETAILED DESCRIPTION:
This is a multi-center, randomized, single-blind*, parallel group, placebo-controlled, study with two dosing regimens in subjects diagnosed with moderate to severe asthma using MN-221 or placebo. Subjects will be randomized to receive MN-221 or placebo in a 3:1 ratio, MN-221:placebo. Subjects randomized to receive MN-221 will be dosed with active study drug at both dosing visits, and subjects randomized to the placebo arm will receive placebo at both dosing visits. Approximately 25 subjects diagnosed with moderate to severe asthma who have not received inhaled corticosteroid therapy within one month of Screen Visit 1 will be enrolled and will participate throughout the study.

Initial dose:

* 16 μg/min for 15 minutes followed by 8 μg/min for 105 minutes (2-hour infusion with a total dose of 1,080 μg MN-221 or Placebo)

Subsequent dose:

* 30 μg/min for 15 minutes followed by 15 μg/min for 45 minutes (1-hr infusion with a total dose of 1,125 μg MN-221 or Placebo)

There will be approximately a two to four week period between each dose regimen, during which time a safety review will be performed before proceeding to the next dose level. Subjects will be screened for eligibility and continued eligibility will be determined for each subject prior to administering each dose. After the initiation of the intravenous infusion of MN-221 or placebo, serial spirometry will be measured for approximately 24 hours.

For each dose evaluation period, subjects will be domiciled in the clinical research unit (CRU) for 2 nights, beginning on Day -1, one day before dosing. Determination of continued study eligibility will be made on Day -1 for each dose level. Day 1 will include study drug infusion and approximately a 24-hour observation period into Day 2 to allow safety monitoring, serial spirometry, and serum PK measurements. Subjects will be discharged from the CRU on Day 2. They will return to the CRU approximately 2-4 weeks later to participate in the subsequent dose group.

*This is a "modified" single-blind study in which the subject and Investigator are both blinded regarding the treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects;
2. Must sign an informed consent;
3. Diagnosis of asthma as defined by the American Thoracic Society for at least 3 months;
4. Must not be receiving inhaled corticosteroids for control within 1 month of study;
5. Must have an increase in FEV1 of at least 12% and 200 cc over the pre-albuterol FEV1 within 30 minutes after inhalation of up to 4 puffs of albuterol via a metered dose inhaler;
6. Non-smoker for at least 6 months and in good health;
7. Female subjects must have a negative pregnancy test;
8. Male and female subjects of child-bearing potential (not surgically sterile or post menopausal) must be abstinent or agree to use contraceptive regimens throughout the study;
9. Subjects receiving allergy desensitization therapy can participate as long as they have been on a stable maintenance dose for ≥ 6 months;
10. Subject must be willing and able not to use inhaled bronchodilators for 6 hours before and until 24 hours after each study drug administration at all study visits; and
11. Subject must demonstrate mental and physical ability and willingness to follow all study-specific instructions pertaining to the scheduling of study visits and assessments.

Exclusion Criteria:

1. Have significant cardiopulmonary, renal, hepatic, endocrine, metabolic, neurological or other systemic disease;
2. Received emergency treatment for asthma within 1 month, or hospitalized for asthma within 3 months;
3. Had an upper or lower respiratory tract infection within 3 weeks, or sinus infection within 7 days;
4. Have participated in a clinical study with an investigational drug, other than an MN-221 study, within 30 days;
5. Have history or evidence of drug or alcohol abuse within 2 years of study entry;
6. Female subjects who are pregnant or lactating;
7. Taking any of the following excluded asthma/allergy medications within the time periods indicated prior to the first study visit:

   * Oral, inhaled, or parenteral corticosteroids for 1 month prior to the first study visit.
   * Anti-IgE medication for 3 months prior to the first study visit.
   * Theophylline, long-acting bronchodilators, and anti-cholinergics for 2 weeks prior to the first study visit.
8. Taking leukotriene modifiers and not on a stable daily dosage for 4 weeks prior to the first study visit.
9. Taking antihistamines, nasal corticosteroids, or decongestants and not on a stable dose for 3 days prior to any dosing day.
10. Have a known allergy to MN-221 or any of the other components of the study drug (i.e. lactose);
11. Have a history of frequent episodes of orthostatic hypotension or any predisposition for orthostatic hypotension;
12. Have used any prescription or over-the-counter medication, vitamin or herbal supplement (except as listed in Inclusion Criterion 7 and Exclusion Criterion 7-10) within 7 days of study entry, or the expected need to use any unapproved prescription or over-the-counter medication or supplement seven days prior to the first study visit until completion of the study;
13. Taking any drugs or substances known to be strong inhibitors of cytochrome P450 enzymes within 10 days of study entry, or the expected need to use such drugs ten days prior to the first study visit until after completion of the study;
14. Taking any drugs or substances known to be strong inducers of cytochrome P450 enzymes within 28 days of study entry, or the expected need to use such drugs prior to completion of the study;
15. Adhering to any special diet that is not well balanced within 28 days of study entry;
16. Have donated (standard donation amount or more) blood or blood products (with the exception of plasma noted below) within 56 days of study entry;
17. Have donated plasma within 7 days of study entry;
18. Have any laboratory value outside the laboratory reference range that is considered to be clinically significant;
19. Have any abnormal vital signs (B/P, respiratory rate, heart rate) considered to be clinically significant;
20. Have positive results for drug and/or alcohol screen;
21. Have any clinically significant ECG abnormality, including a corrected QT interval (QTc) > 450 msec; and/or
22. Have any other medical condition or reason that, in the Investigator's opinion, makes the subject unsuitable to participate in this clinical trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kalafer, Study Director — MediciNova, Inc.
Locations (4):
- United States (4):
  - PRA International, Lenexa, Kansas
  - Northeast Medical Research Associates, North Dartmouth, Massachusetts
  - Clinical Research of the Ozarks, Rolla, Missouri
  - Greenville Pharmaceutical Research, Greenville, South Carolina

REFERENCES:
- [Derived] Matsuda K, Makhay M, Johnson K, Iwaki Y. Evaluation of bedoradrine sulfate (MN-221), a novel, highly selective beta2-adrenergic receptor agonist for the treatment of asthma via intravenous infusion. J Asthma. 2012 Dec;49(10):1071-8. doi: 10.3109/02770903.2012.729631. Epub 2012 Oct 25. PMID 23094708

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects diagnosed with moderate to severe asthma in stable status were recruited at clinic
Pre-assignment Details: Subjects were screened for eligibility and must have demonstrated an improvement in forced expiratory volume in 1 second (FEV1) of at least 12% and 200 cc at the Screen Visit after bronchodilator treatment compared to pre-bronchodilator use. Continued eligibility was determined for each subject prior to administering each dose.
Groups:
- MN-221 1-hour Infusion: 30 μg/min for 15 minutes followed by 15 μg/min for 45 minutes (1-hr infusion with a total dose of 1,125 μg)
- Placebo: MN-221 Placebo continuous infusion
- MN-221 2-hour Infusion: 16 μg/min for 15 minutes + 8 μg/min for 105 minutes (2-hour infusion, total dose 1,080 μg) or placebo
Period: Visit 3/Dose 2
Arm/Group | MN-221 1-hour Infusion | Placebo | MN-221 2-hour Infusion
Started | 10 | 11 | 11
Completed | 9 | 6 | 11
Not Completed | 1 | 5 | 0
Period: Visit 2/Dose 1
Arm/Group | MN-221 1-hour Infusion | Placebo | MN-221 2-hour Infusion
Started | 11 | 6 | 11
Completed | 9 | 5 | 11
Not Completed | 2 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — subject not compliance | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MN-221 1-hour Infusion | Placebo | MN-221 2-hour Infusion | Total
Number analyzed (Participants) | 11 | 6 | 11 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 6 | 11 | 28
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.5 (11.25) | 36.7 (9.65) | 36.7 (9.65) | 32.7 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 13
  Male | 7 | 1 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 11 | 6 | 11 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reported to Have Adverse Events
Time Frame: Day 1 to Day 2
Measure: Number; unit: participants
Arm/Group | MN-221 1-hour Infusion | Placebo | MN-221 2-hour Infusion
Number analyzed (Participants) | 11 | 6 | 11
participants | 11 | 6 | 11

2. Secondary Outcome: FEV1 Percent Predicted Changes From Base Line
Description: The primary efficacy variable will be the change from baseline in FEV1, expressed as percent of predicted at hour 1 after the start of the infusion. Analysis of all other variables at all other time points will be considered secondary.
Time Frame: Day 1 to Day 2
Measure: Mean (Standard Deviation); unit: FEV1 percent predicted
Arm/Group | MN-221 1-hour Infusion | Placebo | MN-221 2-hour Infusion
Number analyzed (Participants) | 11 | 6 | 11
FEV1 percent predicted | 17.48 (10.19) | 1.85 (9.45) | 8.95 (9.2)

ADVERSE EVENTS:
Arm/Group | MN-221 1-hour Infusion | Placebo | MN-221 2-hour Infusion
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/6 | 0/11
Other Adverse Events (participants affected / at risk) | 11/11 | 4/6 | 9/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MN-221 1-hour Infusion (N=11) | Placebo (N=6) | MN-221 2-hour Infusion (N=11)
headache (Nervous system disorders) | 3 (3) | 1 (1) | 2 (3)
tremor (Nervous system disorders) | 5 (5) | 0 (0) | 6 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 4 (4)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram T wave inversion (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Electrocardiogram T wave amplitude decreased (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram ST segment depression (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram QT prolonged (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less